CLINICAL TRIAL: NCT02669043
Title: Physiological and Cognitive Biomarkers for Ketamine's Antidepressant Effects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Assistant in Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015P002397; K23MH107776 (NIH)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine (Experimental): All participants receive open-label ketamine
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Intravenous ketamine 0.5mg/kg over 40 minutes
  Other Names: Ketamine Hydrochloride

SUMMARY:
Anxious depression is a particularly difficult-to-treat subtype of depression. Patients with anxious depression do not respond as well to currently available antidepressant medications. Nevertheless, in previous studies, low dose IV ketamine, which rapidly decreases symptoms of depression within hours in many patients with "treatment-resistant" depression, has been associated with superior efficacy in those individuals with anxious compared with non-anxious depression. In order to understand this unique effect more fully, the current protocol is aimed at further delineating biomarkers of ketamine's effects among individuals with treatment-resistant anxious depression compared to those with nonanxious depression.

ELIGIBILITY:
Inclusion Criteria:

1. be 18-64 years old,
2. read, understand, and provide written informed consent in English,
3. meet criteria for a primary psychiatric diagnosis of Major Depressive Disorder (MDD) for ≥ 4 weeks,
4. have a history ≥1 failed medication trial during the current depression,
5. be on a stable adequate dose of an FDA-approved antidepressant medication for ≥28 days,
6. maintain a treating doctor who is in agreement with study participation,
7. have a reliable chaperone to accompany them home following the completion of the ketamine infusion day,
8. be generally healthy, as assessed by medical history, physical examination (including vital signs), clinical laboratory evaluations, and electrocardiogram (EKG),
9. be of non-childbearing potential or use of an acceptable form of birth control (females only).

Exclusion Criteria:

1. delirium or dementia diagnosis,
2. unstable medical illness or clinically significant laboratory results,
3. history of clinically significant cardiovascular disease or electrocardiogram (EKG) findings, or medical conditions that put the patient at risk for possible cardiac side effects (e.g., requirement of cardiac pacemaker) or alter brain morphology (e.g., recent head trauma, post intracranial surgery, intracranial mass or bleed or unstable sleep apnea), or a blood pressure >140/95 mmHg at Screening,
4. history of multiple adverse drug reactions,
5. current/past history of psychotic disorders, history of out-of-body feelings or derealization,
6. active substance use disorders (except nicotine and caffeine) within the past six months or past history of ketamine/PCP (phencyclidine) abuse (we will confirm this with collateral information from their doctor if necessary),
7. requirement of excluded medications that may interact with ketamine,
8. caffeine or nicotine use within 1 hour of psychophysiology testing, or alcohol use within 1 day of testing,
9. pregnancy, breastfeeding, or unacceptable means of birth control (females only)
10. clinically significant hearing impairment,
11. current serious suicidal or homicidal risk,
12. concurrent participation in other research studies involving medications or other treatments,
13. narrow angle glaucoma,
14. acute intermittent porphyria history,
15. history of seizures in the past 6 months, regardless of seizure type,
16. hyperthyroidism or untreated hypothyroidism,
17. airway instability or pulmonary disease with hypercarbia, or
18. current or past cubital or carpal tunnel syndrome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Ionescu, M.D., Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine
Started | 8
Completed | 4
Not Completed | 4
Not completed — Didn't meet I/E criteria | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48.3 [34 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
HAMD Total Score [Mean (Full Range); unit: units on a scale] — Depression rating scale; possible scores range from 0 to 81 with higher scores indicating higher depression symptoms.
  units on a scale | 28.5 [25 to 31]

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS, HAM-D)
Description: Continuous score of depression symptoms. The higher the score, the more severe the depression. HAMD scores range from 0 to 81.
Time Frame: 48 hours
Population: Patients who completed the study. Outcome measure was at 48 hours.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 4
units on a scale | 11.5 [5 to 27]

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT02669043/Prot_SAP_002.pdf
  • Informed Consent Form (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT02669043/ICF_003.pdf